CLINICAL TRIAL: NCT01365338
Title: Subject And Investigator-Blinded, Sponsor-Open, Randomized, Single-Dose, Placebo-Controlled, Parallel Group Study to Assess Effects of PF-04958242 on Bold Functional MRI During Working Memory Activation and Arterial Spin Labeling at Rest in Healthy Subjects
Brief Title: A Study To Assess Effects Of PF-04958242 On Bold Functional Magnetic Resonance Imaging During Working Memory Activation And Arterial Spin Labeling At Rest In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1701003
Record Dates: First submitted 2011-05-11; First posted 2011-06-03 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo as a single oral dose.
  Interventions: Drug: Placebo
- Cohort 1 (Experimental): Participants will receive 0.075 milligrams (mg) of PF-04958242 as a single oral dose.
  Interventions: Drug: PF-04958242
- Cohort 2 (Experimental): Participants will receive 0.15 mg of PF-04958242 as a single oral dose.
  Interventions: Drug: PF-04958242

INTERVENTIONS:
Drug: Placebo — Administered as specified in the treatment arm
  Arms: Placebo
Drug: PF-04958242 — Administered as specified in the treatment arm
  Arms: Cohort 1; Cohort 2

SUMMARY:
The primary objective of this study aims to determine whether the drug affects brain activity in healthy volunteers, either when the participants are performing a memory task, or when lying at rest. Subjects will undergo a brain scan under both of these conditions after a dose of either the study drug or a placebo is administered.The secondary objective is to evaluate the safety and tolerability of the four doses of PF-04958242 administered orally to healthy adult participants.

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Body Mass Index (BMI) of 17.5 to 30.5 kilograms per meter squared (kg/m2);
* Total body weight >50 kilograms (kg) (110 pounds [lbs]);

Key Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing);
* Positive urine drug screen;
* Pregnant or nursing females, and females of child bearing potential;
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2011-06-24 (Actual); Primary Completion 2012-12-14 (Actual); Study Completion 2012-12-14 (Actual)

PRIMARY OUTCOMES:
Functional Magnetic Resonance Imaging Data During Working Memory Task | 59 Minutes Post-dose
Arterial Spin Labeling Data | 39 Minutes Post-dose

SECONDARY OUTCOMES:
Number of Participants Experiencing Adverse Events and Serious Adverse Events | Up to Day 11
  An adverse event is any untoward medical occurrence in a clinical investigation participant administered a product or medical device. A serious adverse event or serious adverse drug reaction is any untoward medical occurrence at any dose that: Results in death; Is life-threatening (immediate risk of death); Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent or significant disability/incapacity; Results in congenital anomaly/birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, New Haven, Connecticut, United States